CLINICAL TRIAL: NCT03888534
Title: Open-Label Phase 1 Study to Assess the Maximum Tolerated Dose, Pharmacokinetics, and Safety of Ixazomib Administered Intravenously to Pediatric Patients Aged 0 to <18 Years With Relapsed or Refractory Acute Lymphoblastic Leukemia, With or Without Extramedullary Disease, or Relapsed or Refractory Lymphoblastic Lymphoma
Brief Title: Intravenous Ixazomib in Pediatric Participants With Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL) or Lymphoblastic Lymphoma (LLy)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision (no safety or efficacy concerns)
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C16051; U1111-1225-3528 (Registry Identifier: WHO); 2018-003907-20 (EudraCT Number)
Record Dates: First submitted 2019-03-22; First posted 2019-03-25 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Ixazomib, injection, intravenously, once on Days 1, 4, 8, and 11 in a single 29-day treatment cycle in combination with multiagent reinduction therapy. Participants >= 1 year will receive the starting dose of 1.0 milligram per square meter (mg/m^2) and <1 year will receive the starting dose of 0.03 milligram per kilogram (mg/kg). The dose escalation phase will determine the MTD or RP2D of Ixazomib. Dose of Ixazomib will be escalated based on the observed safety and tolerability data.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib intravenous injection in combination with reduction chemotherapy.
  Other Names: MLN9708

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D), safety and toxicity, and pharmacokinetics (PK) of ixazomib administered intravenously in combination with multiagent reinduction chemotherapy in pediatric participants with relapsed/refractory ALL or LLy.

DETAILED DESCRIPTION:
29-Apr-2020 Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

The drug being tested in this study is called Ixazomib. Ixazomib is being tested to determine the MTD or RP2D of intravenous ixazomib when administered in combination with multiagent chemotherapy (reinduction therapy) in pediatric participants with relapsed or refractory ALL or relapsed/refractory LLy.

The study will enroll approximately 18 participants. Doses of ixazomib will be escalated according to a standard 3+3 dose escalation schema. Participants aged >= 1 year will receive the starting dose of 1.0 mg/m^2 and participants aged <1 year will receive the starting dose of 0.03 mg/kg. Ixazomib will be administered in combination with multiagent reinduction therapy. The dose escalation phase will determine the MTD and/or RP2D of ixazomib. Dose escalation will be based on the observed safety and tolerability data.

Participants aged <1 year will be assessed separately and will not contribute to the dose escalation assessment.

This multi-center trial will be conducted in the United States and Spain. The overall time to participate in this study is approximately 30 months. Participants will be followed up to Day 60 after the first dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed/refractory ALL with or without extramedullary disease, including central nervous system (CNS)2 (<5 white blood cell [WBC]/mcL] in the cerebrospinal fluid [CSF] with blasts) and CNS3 (>=5 WBC/mcL in the CSF with blasts), or relapsed/refractory LLy. Participants with mixed-phenotype ALL or mature (Burkitt-like) leukemia are excluded.
2. Relapsed/refractory ALL must have >=5% blasts in the bone marrow by morphology.
3. Relapsed/refractory LLy participants must have measurable disease documented by clinical, radiologic, and histologic criteria.
4. A Karnofsky performance status of >=50% (for participants aged >16 years) and a Lansky performance status of >=50% (for participants aged <=16 years).
5. Adequate organ function.
6. Failure of 1 or more therapeutic attempts.
7. Full recovery from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy before entering this study, as follows:

   * Cytoreduction with hydroxyurea: Hydroxyurea can be initiated and continued for up to 24 hours before the start of protocol therapy.
   * Cytotoxic therapy: At least 14 days must have elapsed since the completion of the last dose of chemotherapy, except intrathecal (IT) chemotherapy and/or maintenance therapy, such as vincristine (VCR), mercaptopurine, methotrexate, or glucocorticoids. There is no waiting period for those relapsing on maintenance therapy.
   * Hematopoietic stem cell transplantation (HSCT): Participants who have relapsed after HSCT are eligible, provided they have no evidence of acute or chronic graft-versus-host disease (GVHD), are not receiving GVHD prophylaxis or treatment, and are at least 90 days posttransplant at the time of enrollment.
   * Hematopoietic growth factors: At least 7 days must have elapsed since the completion of therapy with granulocyte colony-stimulating factor (G-CSF) or other growth factor at the time of enrollment. At least 14 days must have elapsed since the completion of therapy with pegfilgrastim.
   * Biologic (antineoplastic agent): At least 7 days must have elapsed since the last dose of a biologic agent. For agents that have known adverse events (AEs) occurring beyond 7 days after the end of administration, this period must be extended beyond the time during which AE are known to occur. The duration of this interval must be approved by the project clinician (or designee).
   * Monoclonal antibodies: At least 3 half-lives must have elapsed after the last dose of an administered monoclonal antibody.
   * Immunotherapy: At least 30 days must have elapsed after the completion of any type of immunotherapy (example, tumor vaccines, chimeric antigen receptor T-cells).
   * Photon radiotherapy (XRT): Craniospinal XRT is prohibited during protocol therapy. No washout period is necessary for radiation given to any extramedullary site other than the CNS; >=90 days must have elapsed if prior total body irradiation or craniospinal XRT was given.
   * Anthracyclines: Participants must have had a lifetime exposure of <400 mg/m^2 of doxorubicin equivalents of anthracyclines.
   * Proteasome inhibitors: Participants with a prior exposure to proteasome inhibitor (PIs) (example, bortezomib, carfilzomib) are eligible as long as the participant demonstrated at least a partial response to chemotherapy with a PI.

Exclusion criteria:

1. ALL participants: have isolated extramedullary disease, including CNS or testicular disease.
2. Have Grade >=2 peripheral sensory or motor neuropathy, defined by the Modified "Balis" Pediatric Scale of Pediatric Neuropathies, at the time of enrollment.
3. Have a planned administration of chemotherapy, radiation therapy, or immunotherapy, other than the study drugs used for this protocol.
4. Have deoxyribonucleic acid fragility syndromes (example, Fanconi anemia, Bloom syndrome).
5. Have Down syndrome.
6. Are receiving cyclosporine, tacrolimus, or other agents to prevent graft-versus host disease (GVHD) after HSCT.
7. Have Philadelphia chromosome (Ph)-positive ALL or Ph-like ALL and are currently receiving tyrosine kinase inhibitor therapy.
8. Are receiving systemic treatment with strong inducers of cytochrome P450 3A (CYP3A)(example,rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital, St. John's wort) within 14 days before study enrollment.
9. Are receiving systemic treatment with strong CYP3A inhibitors within 14 days before study enrollment.
10. Are receiving systemic treatment with inhibitors or inducers of P-glycoprotein (P-gp) within 14 days before study enrollment.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLT) During Reinduction Chemotherapy | Up to Day 29
  DLT: Grade 4 nonhematologic toxicity after first dose of ixazomib and is probably/definitely attributable to the ixazomib treatment regimen, with exceptions, example fever/infection with/without hospitalization, fatigue and gastrointestinal symptoms, hypofibrinogenemia, metabolic/laboratory abnormalities that resolve to less than or equal to(<=)Grade 2 within 7 days. Any Grade 3/4 nonhematologic toxicity after first dose of ixazomib that is possibly/probably/definitely attributable to the ixazomib treatment regimen and results in omission of subsequent dose of chemotherapy, with exception of fever/infection. Hematologic toxicities: Failure to recover a peripheral absolute neutrophil count (ANC) ≥0.5*10^9 per liter (/L) and a platelet count ≥50*10^9/L due to documented bone marrow hypoplasia (cellularity <10 20%) within 42 days after the beginning of systemic chemotherapy without evidence of active disease by bone marrow evaluation or active infection.
Number of Participants With Grade 3 or Higher Treatment Emergent Adverse Events (TEAEs) Based on Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | Up to 30 months
Number of Participants With Worst Shift From Baseline Values to Post-baseline Values in Clinical Laboratory Parameters | Up to 30 months
AUCt: Area Under the Plasma Concentration-time Curve From Time 0 to Time t for Ixazomib | Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose and Day 11 pre-dose and at multiple time points (up to 264 hours) post-dose
Cmax: Maximum Observed Plasma Concentration for Ixazomib | Day 1 pre-dose and at multiple time points (up to 72 hours) post-dose and Day 11 pre-dose and at multiple time points (up to 264 hours) post-dose

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 30 months
  ORR is defined as the percentage of participants with complete response (CR) or CR with incomplete platelet recovery (CRp) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR is defined as bone marrow with less than 5 percent (%) blast by morphology, no evidence of circulating blasts or extramedullary disease, and recovery of peripheral counts (ANC >=1.0*10^9/L and a platelet count >=100*10^9/L). CRp is defined as bone marrow with <5% blasts by morphology, no evidence of circulating blasts or extramedullary disease, and recovery of ANC (>1000/mcL) but insufficient recovery of platelets (counts <100, 000/mcL).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (4):
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - St Jude Children's Research Hospital, Memphis, Tennessee
- Spain (3):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - C.H. Regional Reina Sofia, Córdoba
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.